CLINICAL TRIAL: NCT05629949
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Phase III Study of the Efficacy and Safety of QL1701 Plus Docetaxel Versus Herceptin® Plus Docetaxel as First Line Therapy in Patients With HER2-positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1701-002
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1701+Docetaxel (Experimental): Participants received intravenous infusion of QL1701 with docetaxel. The initial load dose of QL1701 was 8mg/kg, followed by 6mg/kg every three weeks; The recommended dose of docetaxel is 75mg/m2, given once every 3 weeks for a treatment cycle of 3 weeks.
  Interventions: Drug: QL1701; Drug: Docetaxel
- Herceptin®+Docetaxel (Active Comparator): Participants received intravenous infusion of Herceptin® with docetaxel. The initial load dose of Herceptin® was 8mg/kg, followed by 6mg/kg every three weeks; The recommended dose of docetaxel is 75mg/m2, given once every 3 weeks for a treatment cycle of 3 weeks.
  Interventions: Drug: Herceptin®; Drug: Docetaxel

INTERVENTIONS:
Drug: QL1701 — 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles.
  Arms: QL1701+Docetaxel
Drug: Herceptin® — 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles.
  Arms: Herceptin®+Docetaxel
Drug: Docetaxel — The recommended dose is 75mg/m2 and the infusion time is approximately 70min (±20min) (or adjusted according to clinical experience at each study center). The drug was administered once every 3 weeks for a treatment cycle of 3 weeks, with the exception of the second day of the first cycle, followed by the first day of each cycle for at least 8 cycles

SUMMARY:
This is a Phase III, double-blind, randomized multicenter study to compare the efficacy and to evaluate the safety and immunogenicity of QL1701 and Herceptin® in patients with human epidermal growth factor receptor 2 (HER2)-positive, locally recurrent or previously untreated metastatic breast cancer.

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomized multicenter study to compare the efficacy and to evaluate the safety and immunogenicity of QL1701 and Herceptin® in patients with human epidermal growth factor receptor 2 (HER2)-positive, recurrent or previously untreated metastatic breast cancer. Eligible patients will be assessed centrally for HER2 status and the presence of at least one measurable target lesion before randomization. Patients will undergo a tumor assessment for evaluation of response according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) every 6 weeks up to 24 weeks (regardless of the number of cycles actually given);

ELIGIBILITY:
Inclusion Criteria:

1. Patients have voluntarily agreed to participate and given written informed consent.
2. Female ≥18 years of age on day of signing the informed consent form (ICF).
3. Histologically or cytologically confirmed adenocarcinoma of the breast that is HER2-positive by molecular pathology [IHC or fluorescence in situ hybridization (FISH)]; (4) Locally recurrent or metastatic breast cancer (including patients with first diagnosis of metastatic breast cancer) that cannot be treated with radical surgery or radiotherapy has an indication of taxane antitumor drug therapy regimen (according to the NCCN or Chinese treatment guidelines); (5) No systemic chemotherapy or targeted drug therapy for metastatic breast cancer has been performed in the past. If endocrine therapy has been performed, it must be stopped at least 2 weeks before enrollment; For patients who had received relevant neoadjuvant or adjuvant therapy in the past, HER2- related drugs should have been discontinued for at least 12 months before enrollment, and other non-HER2-related drugs should have been discontinued for at least 1 month before enrollment.

   * There is at least one measurable lesion (non-bone metastatic lesion), which was evaluated according to RECIST 1.1 criteria.

Exclusion Criteria:

1. Previous systemic chemotherapy or targeted drug therapy for metastatic breast cancer (including Herceptin ®, such as trastuzumab, pertuzumab, TDM-1, etc.; And non-herceptin ®, such as lapatinib, pyrrotinib, neratinib, etc.);
2. Currently receiving other systemic antitumor therapies (such as chemotherapy and/or immunotherapy) or other therapies not specified in the study protocol that may affect the study;
3. Use of other investigational drugs within 28 days before signing the informed consent;
4. Definite confirmation of brain metastases (except those that have been evaluated asymptomatic or asymptomatic for at least 4 weeks after local lesion management and do not require steroid treatment);
5. Have a history of other malignant tumors within 5 years before signing the informed consent, excluding cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has received radical treatment;

   * Previous HIV infection or HIV screening positive, or HCV RNA positive, or syphilis antibody positive and active titer test;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
ORR at Week 24 by IRC | From time of First treatment to week 24
  calculated as the proportion of patients with a best response of complete response (CR) or partial response (PR) from first assessment until Week 24 according to RECIST 1.1.

SECONDARY OUTCOMES:
ORR at Week 24 by Investigator | From time of First treatment to week 24
  alculated as the proportion of patients with a best response of complete response (CR) or partial response (PR) from first assessment until Week 24 according to RECIST 1.1.
PFS up to 12 months | From time of first treatment to 12 months
  The probability of being alive without documented progression up to 12 months after randomization
DoR | From time of first treatment to 12 months
  The time from first documentation of CR or PR to the first documentation of progression
DCR | From time of first treatment to 12 months
  The proportion of patients who achieve CR, PR, or stable disease (SD) of at least 12 weeks
Overall survival at 12 months | From time of first treatment to 12 months
  the probability of being alive 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital,Chinese Academy of Medical Sciences, Beijing, China